CLINICAL TRIAL: NCT06058754
Title: Evaluating Group-based (ADAPT) Versus One-to-one (Usual) Occupational Therapy on Ability to Perform Activities of Daily Living (ADL) in People With Chronic Conditions (Go:OT Trial)
Brief Title: Group-based [ADAPT] Versus One-to-one [Usual] Occupational Therapy (Go:OT Trial)
Acronym: Go:OT
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Parker Research Institute (Other)
Collaborators: Rehabilitation Center Rødovre Municipality (Genoptræning Rødovre Kommune) (Unknown); Den Kommunale Kvalitetsudviklingspulje (Unknown); Lundbeckpuljen (Unknown); Oak Foundation (Other); Tværspuljen (Unknown)
Responsible Party: Principal Investigator, Eva Ejlersen Wæhrens, Senior researcher, Associate Professor, Parker Research Institute
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Health Services Research
Other Study IDs: Parker Institute,
Record Dates: First submitted 2023-09-15; First posted 2023-09-28 (Actual); Last update posted 2023-09-28 (Actual); Status verified 2023-09

CONDITIONS: Chronic Condition; Chronic Disease; Chronic Conditions, Multiple
Keywords: Occupational therapy; ADL; Adaptation; Chronic condition; Peer-exchange; group-based
MeSH Terms: conditions — Chronic Disease; Multiple Chronic Conditions | interventions — Acclimatization; Occupational Therapy

STUDY DESIGN:
Intervention Model Description: A single-center, double-blinded, randomized, parallel-group, equivalence 6-months follow-up study with external pilot, effect, process and economic evaluations
Who Masked: Participant, Outcomes Assessor
Masking Description: Participants are informed that they will be allocated to one of two occupational therapy intervention programs that both aims to improve ADL ability, but overall primarily differ in terms of their format i.e. a group-based versus a one-to-one intervention program format. Participants are not informed, which of the two types of formats that are the new experimental intervention format (ADAPT) nor control (UOT). Baseline assessments are conducted prior to randomization by a local employed occupational therapists, who is instructed not to reveal which intervention that is the new experimental intervention. The post and follow-up assessors, a research occupational therapy assistant employed at the Parker Institute, is also instructed not to disclose which intervention that is the new experimental one. Finally, all participants are reminded not to disclose any details, that may provide the outcome assessors with insights regarding their allocated study arm.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ADAPT Program (Experimental): The ADAPT Program is a structured and individualized group-based program
  Interventions: Behavioral: The ADAPT Program
- Usual Occupational Therapy (UOT) (Active Comparator): UOT is delivered by one occupational therapist in the clients homes or local environments. .
  Interventions: Behavioral: UOT

INTERVENTIONS:
Behavioral: The ADAPT Program — The ADAPT Program is a structured and individualized 10-week group-based program, in which two occupational therapists teach groups of people, the skills of problem-solving more efficiently as means to overcome ADL task performance problems. The ADAPT Program 3.0 includes 2 individual two-hour sessions (sessions 1 and 10) conducted in the clients homes and eight two-hour group-based sessions (sessions 2-9). Moreover, two booster sessions (sessions 11 and 12) are delivered to support sustainable gains after termination of the 10-week ADAPT Program 3.0
  Other Names: Adaptation; Compensatory; occupational therapy; group-based; peer-exchange; problem-solving
  Arms: ADAPT Program
Behavioral: UOT — UOT is delivered by one occupational therapist. Sessions are individualised and focused on improving ADL ability e.g. by practicing the performance of ADL task or adjusting home environments. UOT typically includes 7 one-to-one sessions of 60 minutes, delivered over a 10-week period in the clients´ homes. The dose is however not fixed but based on the occupational therapists´ clinical judgement in collaboration with the individual client
  Other Names: Usual occupational therapy
  Arms: Usual Occupational Therapy (UOT)

SUMMARY:
This trial aims to evaluate the ADAPT Program in terms of efficacy, process and cost-efficacy compared to usual occupational therapy (UOT) in people with decreased ability to perform activities of daily living (ADL) following chronic conditions. As both the ADAPT Program and UOT are targeted improvements in ADL ability, the primary objective of this trial is to assess equivalence between the ADAPT Program and UOT on changes in ADL ability as measured with the Assessment of Motor and Process Skills (AMPS).

DETAILED DESCRIPTION:
Background: The number of people living with chronic conditions limiting the ability to perform activities of daily living (ADL) tasks is increasing. Occupational therapists are trained to deliver interventions to improve ADL ability, e.g. by adapting and adjusting daily routines and physical environments. Municipality occupational therapy (OT) interventions are usually delivered as one-to-one sessions in the client´s home. While this intervention format might be effective in improving ADL ability, a group-based intervention format might be as effective but more cost-effective and hold other secondary gains. Guided by the British Medical Research Council's guidance (MRC) on how to develop and evaluate complex interventions, the ADAPT Program, a peer-exchange group-based program, was developed, piloted, and evaluated for its functioning and feasibility in municipality settings. These studies provided initial evidence for the ADAPT Programs effectiveness in improving ADL ability and suggests gains as improved well-being. Hence, the current phase concerns a full-scale evaluation of the ADAPT Program including evaluation of effectiveness, processes and cost-effectiveness.

Material and Methods: The randomized controlled trial (RCT), initiated with an external pilot (n=12), will include 130 home dwelling persons with decreased ADL ability following chronic conditions. Participants are randomized to either ADAPT Program (experimental) or usual OT (control).

Primary outcome: Observed ADL motor ability measured with the Assessment of Motor and Process Skills (AMPS).

Secondary outcomes: Observed ADL process ability measured with the AMPS; patient reported ADL task Performance and Satisfaction measured with the ADL-Interview (ADL-I, Performance and Satisfaction scores); Well-being assessed with the World Health Organisation-Five Well Being Index (WHO-5); Health-related Quality of Life assessed with the European Quality of Life - 5 Dimensions (EQ-5D).

Exploratory outcomes include patient reported changes, using transition scales to evaluate participants´ experience of a) changed ADL task performance and satisfaction, b) changed problem-solving skills, c) changed quality of life, d) changed global health, e) changed needs for assistance. Finally, participants are to rate their overall experience of the allocated occupational therapy intervention.

Data collection: Effectiveness and cost-effectiveness data are collected at baseline and post intervention i.e., 3-months (week 12) and 6-months (week 26) from baseline. Costs will be estimated based on micro costing and national registries. Effects will be Quality Adjusted Life Years and changes in AMPS ADL motor ability. Process evaluation data will be collected using registration forms and semi-structured qualitative interviews.

ELIGIBILITY:
Inclusion criteria:

* ≥ one year since medical diagnosed with one or more chronic conditions.
* Lives in own home.
* Experience ADL task performance problems.
* Show ADL motor ability measures <1.50 logits on the AMPS ADL motor skill scale (indicate increased effort during ADL task performance).
* Communicate independently and relevantly orally and in writing.
* Willing and interested in attending occupational therapy interventions focused on improving ADL task performance.

Exclusion criteria:

* ADL process ability measures <0.00 indicating that the person is unlikely to profit from educational programs focused on using adaptational strategies.
* Personal ADL (PADL) problems with acute need for help.
* Mental illness and/or other acute (<3 months) conditions effecting ADL task performance significantly.
* Significant communication barriers (significant cognitive deficits, -aphasia, -hearing loss, -dyslexia and/or -language barriers).
* Known substance abuse.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 130 (Estimated)
Dates: Start 2023-09-04 (Actual); Primary Completion 2024-09-27 (Estimated); Study Completion 2024-12-06 (Estimated)

PRIMARY OUTCOMES:
Change in observed ADL motor ability, Assessment of Motor and Process Skills (AMPS) | week 12
  Observation-based ADL motor ability (reflecting physical effort and independence ). Linear measures of ADL motor ability generated using Rasch measurement models. Higher scores mean better ADL ability

SECONDARY OUTCOMES:
Change in observed ADL motor ability, using AMPS | week 26
  Observation-based ADL motor ability (reflecting physical effort and independence ). Linear measures of ADL motor ability generated using Rasch measurement models. Higher scores mean better ADL ability
Change in observed ADL process ability, using AMPS | week 12
  Observation-based ADL process ability (reflecting efficiency, safety and independence). Linear measures of ADL process ability generated using Rasch measurement models. Higher scores mean better ADL ability
Change in observed ADL process ability, using AMPS | week 26
  Observation-based ADL process ability (reflecting efficiency, safety and independence). Linear measures of ADL process ability generated using Rasch measurement models. Higher scores mean better ADL ability
Change in self-reported ADL ability, using the ADL-Interview (ADL-I), Performance scale | week 12
  Self-reported ability to perform ADL tasks, based on interview. Linear measures of ADL ability generated using Rasch measurement models. Higher scores mean better ADL ability
Change in self-reported ADL ability with ADL-I, Performance scale | week 26
  Self-reported ability ot perform ADL tasks, based on interview. Linear measures of ADL ability generated using Rasch measurement models. Higher scores mean better ADL ability
Change in self-reported satisfaction with ADL ability, using ADL-I, Satisfaction scale | week 12
  Self-reported satisfaction with ADL task performance, based on interview. Linear measures of ADL ability generated using Rasch measurement models. Higher scores means higher satisfaction
Change in self-reported satisfaction with ADL ability, using the ADL-Interview (ADL-I), Satisfaction scale | week 26
  Self-reported satisfaction with ADL task performance, based on interview. Linear measures of ADL ability will be generated using Rasch measurement models. Higher scores means higher satisfaction
Well-being, using the World Health Organisation- Five Well-Being Index (WHO-5) | week 12
  Participants are asked to rate well being in regard to five questions. Response options are scored on a 6-point scale in which 0=at no time to 0=all the time. Lower scores are lower well-being
Well-being, using The World Health Organisation- Five Well-Being Index (WHO-5) | week 26
  Participants are asked to rate well being in regard to five questions. Response options are scored on a 6-point scale in which 0=at no time to 0=all the time. Lower scores are lower well-being
Quality of life, using the EuroQoL 5 dimensions (EQ-5D) | week 12
  Participants are asked to rate 5 aspects of health-related quality of life Quality of life in regard to five items scores on a 5 point likert scale from I am not/have none to I have extreme/i cannot
Quality of life, using EQ-5D | week 26
  Participants are asked to rate 5 aspects of health-related quality of life Quality of life in regard to five items scores on a 5 point likert scale from I am not/have none to I have extreme/i cannot

OTHER OUTCOMES:
Perceived change in ADL task performance, TRANS-Questionnaire | week 12
  Participants are asked about their experienced change in a) performance of ADL tasks and b) satisfaction witt their ADL ability following occupational therapy intervention. Response options are scored on a 7-point likert scale from 'markedly worse' to 'markedly better'
Perceived change in ADL task performance, TRANS-Questionnaire | week 26
  Participants are asked about their experienced change in a) performance of ADL tasks and b) satisfaction witt their ADL ability following occupational therapy intervention. Response options are scored on a 7-point likert scale from 'markedly worse' to 'markedly better'
Perceived change in problem-solving skills, TRANS-Questionnaire | week 12
  Participants are asked about their experienced change in a) identifying daily task performance problems and b) the ability to solve task performance problems following occupational therapy intervention. Response options are scored on a 7-point likert scale from 'markedly worsened' to 'markedly better'
Perceived change in problem-solving skills, TRANS-Questionnaire | week 26
  Participants are asked about their experienced change in a) identifying daily task performance problems and b) the ability to solve task performance problems following occupational therapy intervention. Response options are scored on a 7-point likert scale from 'markedly worsened' to 'markedly better'
Perceived change in Quality of Life, TRANS-Questionnaire | week 12
  Participants are asked about their experienced change in a) overall functioning, b) mental well-being, c) physical well-being and d) social well-being following occupational therapy intervention. Response options are scored on a 7-point likert scale from 'markedly bigger' to 'markedly less'
Perceived change in Quality of Life, TRANS-Questionnaire | week 26
  Participants are asked about their experienced change in a) overall functioning, b) mental well-being, c) physical well-being and d) social well-being following occupational therapy intervention. Response options are scored on a 7-point likert scale from 'markedly bigger' to 'markedly less'
Perceived change in global health, TRANS-Questionnaire | week 12
  Participants are asked about their experienced change in global health following occupational therapy intervention. Response options are scored on a 7-point likert scale from 'markedly worse' to 'markedly better'
Perceived change in global health, TRANS-Questionnaire | week 26
  Participants are asked about their experienced change in global health following occupational therapy intervention. Response options are scored on a 7-point likert scale from 'markedly worse' to 'markedly better'
Perceived change in assistance needed, TRANS-Questionnaire | week 12
  Participants are asked about their experienced change in needing assistance in a) findings ways to ease task performance, b) accepting my chronic condition, c) managing symptoms following occupational therapy intervention. Response options are scored on a 7-point likert scale from 'markedly bigger' to 'markedly less'
Perceived change in assistance needed, TRANS-Questionnaire | week 26
  Participants are asked about their experienced change in needing assistance in a) findings ways to ease task performance, b) accepting my chronic condition, c) managing symptoms following occupational therapy intervention. Response options are scored on a 7-point likert scale from 'markedly bigger' to 'markedly less' less
Overall experience of the occupational therapy intervention | week 12
  Participants are asked to rate their experience on a 5 point Likert scale ranging from "excellent' to 'very poor'

CONTACTS AND LOCATIONS:
Overall Officials: Cecilie von Bülow, PhD, Principal Investigator — Parker Institute, Bispebjerg and Frederiksberg Hospital
Locations (1):
- The Parker Research Institute, Department of Rheumatology, Copenhagen University Hospital, Bispebjerg and Frederiksberg Frederiksberg, Denmark, Frederiksberg, Denmark